CLINICAL TRIAL: NCT05980364
Title: In Cardiac Rehabilitation The Effect of Technology-Based Education Structured According to the Health Promotion Model on Healthy Lifestyle Behaviors, Health Fatalism and Risk Knowledge Level: A Randomized Controlled Study
Brief Title: Cardiac Rehabilitation in Coronary Artery Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice Karabulak (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Hatice Karabulak, PhD student, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 02/60
Record Dates: First submitted 2023-07-29; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Have a Diagnosis of Coronary Artery Disease
Keywords: Nursing; cardiac rehabilitation; health promotion model; healthy lifestyle behaviors; health fatalism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Other: Technology-based training structured according to the Health Promotion Model
- Control group (No Intervention)

INTERVENTIONS:
Other: Technology-based training structured according to the Health Promotion Model — Experimental group: A video recording was created with a total of 6 zoom applications to be shared with the patients. The content of the video recordings consists of a presentation accompanied by a slide show with open-ended questions prepared by considering the basic concepts of the trainings and the Health Promotion Model. Video recordings, each of which lasted approximately 15-25 minutes, were shared with patients once a week for a total of 6 weeks via WhatsApp. After each video, patients were given three days to watch the video recordings and create their own responses. After this three-day period, the researcher called the patients with whom he shared the content and gave counseling for 10-15 minutes and received feedback. Follow-up was done in the second 6-week period. During the monitoring process, two reminder interviews were made over the phone, with an interval of 2 weeks, for reminder and counseling, and the post-test data were collected at the end of the monitoring period.
  Arms: Experimental group

SUMMARY:
Cardiac rehabilitation is approaches that focus on accelerating the recovery process of patients after a cardiac event, improving their physical, psychological and social conditions, and controlling risk factors. Cardiac rehabilitation is known to be an effective and cost-effective approach in the secondary prevention of cardiovascular diseases, most of which are caused by preventable risks. Ischemic heart diseases, one of the cardiovascular diseases, are responsible for 16% of total deaths in the world and have increased significantly since 2000, causing 8.9 million deaths in 2019.

When coronary artery diseases cannot be prevented, the basic approach should be to ensure the individual's compliance with treatment and healthy lifestyle behaviors, and to increase the quality of life and life span.

For this reason, the aim of the study is to examine the effects of technology-based education structured according to the health promotion model in cardiac rehabilitation on healthy lifestyle behaviors, health fatalism and risk knowledge level.

Question 1. Does technology-based education structured according to the health promotion model affect the healthy lifestyle behaviors score? Question 2. Does technology-based education structured according to the health promotion model affect the health fatalism score? Question 3. Does technology-based education structured according to the health promotion model affect the cardiovascular disease risk factors knowledge level score?

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of coronary artery disease (acute coronary syndrome, coronary revascularization, atherosclerotic heart disease, etc.),
* Being stable in health (the patient's health status does not change suddenly and is under control),
* If an interventional procedure has been performed, at least three months have passed after discharge,
* Being between the ages of 18-65,
* Being literate,
* Using smart phone and internet,
* Living in the city center

Exclusion Criteria:

* Having a disability (vision, hearing, neurological, cognitive, etc.) that may interfere with education,
* Cardiac rehabilitation is contraindicated
* To have participated in a cardiac rehabilitation program given by another institution before or during the study,

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Change in healthy lifestyle behaviors score | 12 weeks
  Increase in healthy lifestyle behaviors score
Change in health fatalism score | 12 weeks
  Decrease in health fatalism score
Change in cardiovascular disease risk knowledge level score | 12 weeks
  Increase in cardiovascular disease risk knowledge level score

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr.Canturk Capik, Study Director — Ataturk University, Department of Public Health Nursing
Locations (1):
- Kars Harakani State Hospital, Kars, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No